CLINICAL TRIAL: NCT02588521
Title: A Randomized, Double-blind, Placebo-controlled, First-in-human, Study of Orally Administered AL-794 to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single and Multiple Ascending Doses, and the Antiviral Activity of Multiple Doses in an Influenza Challenge Study in Healthy Subjects
Brief Title: A Study of AL-794 to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single and Multiple Doses, and the Antiviral Activity of Multiple Doses in an Influenza Challenge Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alios Biopharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AL-794-801
Record Dates: First submitted 2015-10-14; First posted 2015-10-28 (Estimated); Last update posted 2017-10-11 (Actual); Status verified 2017-10

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — sfericase

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (2):
- AL-794 (Experimental): AL-794 administered orally in a suspension
  Interventions: Drug: AL-794
- Vehicle (Placebo Comparator): Suspension vehicle alone
  Interventions: Other: Placebo/Vehicle

INTERVENTIONS:
Drug: AL-794
  Arms: AL-794
Other: Placebo/Vehicle — Suspension vehicle without active drug
  Arms: Vehicle

SUMMARY:
This randomized, double-blind, placebo-controlled, 4 part study will assess the safety, tolerability, pharmacokinetics and antiviral activity of orally administered AL-794 in healthy volunteers (HV).

ELIGIBILITY:
Inclusion Criteria:

1. Subject has provided written consent.
2. In the investigator's opinion, the subject is able to understand and comply with protocol requirements, instructions, and protocol stated restrictions and is likely to complete the study as planned.
3. Subject is in good health as deemed by the investigator, based on the findings of a medical evaluation including medical history, physical examination, laboratory tests and ECG.
4. Male or female, 18-60 years of age (Parts 1-3). For Part 4, Males or female, 18-55 years of age.
5. Body mass index (BMI) 18-30kg/m2, inclusive. The minimum weight is 50 kg.
6. A female subject is eligible to participate in this study if she is of non childbearing potential or postmenopausal and not receiving hormone replacement therapy.
7. If male, subject is surgically sterile or practicing specific forms of birth control until 90 days after the end of the study.

Exclusion Criteria:

1. Clinically significant cardiovascular, respiratory, renal, gastrointestinal, hepatic, hematologic, neurologic, thyroid or any other medical illness or psychiatric disorder, as determined by the Investigator, and/or Sponsor's Medical Monitor.
2. Positive screening test for hepatitis A, B, C or HIV infection.
3. Clinically significant laboratory abnormalities or abnormalities which are deemed to interfere with the ability to interpret study data.
4. Creatinine clearance of less than 60 mL/min (Cockroft Gault).
5. Total bilirubin, ALT, AST, or Alkaline Phosphatase > 1.2 X ULN.
6. Any condition that, in the opinion of the investigator, would compromise the study's objectives or the well-being of the subject or prevent the subject from meeting the study requirements.
7. Participation in an investigational drug trial or having received an investigational vaccine within 3 months prior to study medication (or inoculation for Part 4 subjects).
8. Clinically significant abnormal ECG findings.
9. Clinically significant blood loss or elective blood donation of significant volume (i.e., > 500 mL) within 90 days of first dose of study drug
10. Heart rate, respiratory rate, temperature or blood pressure values outside of the normal range, per local standards.
11. Unwilling to abstain from alcohol for 1 week before the start of admission until the final Completion Visit assessments.
12. History of regular alcohol intake > 14 units per week of alcohol for females and > 21 units per week for males (one unit is defined as 8 g alcohol) within 3 months of admission.
13. For Parts 1-3, subjects with a history of tobacco use or use of nicotine-containing products within 2 weeks of the screening visit. For Part 4, subjects who have a significant history of any tobacco use at any time.
14. The subject has a positive pre-study drug screen.
15. The use of concomitant medications, including prescription, over the counter medications, herbal medications, inducers or inhibitors of CYP450 enzymes or drug transporters (including P-gp), within 14 days prior to the first dose of study medication, unless approved by the Sponsor's Medical Monitor. Occasional use of ibuprofen or acetaminophen is permitted.
16. Exposure to more than four new investigational entities within 12 months prior to the first dosing day (Parts 1-3) or inoculation (Part 4).
17. Evidence of active infection, including respiratory tract infection within 2 weeks prior to admission.
18. Pregnant or nursing females, or women of childbearing potential. Men whose female partners are pregnant or contemplating pregnancy from the date of screening until 90 days after end of study.
19. Hypersensitivity to the active substances or to any of the excipients of AL-794.
20. Unwillingness or inability to comply with the study protocol for any other reason.
21. Part 4 ONLY: Contraindications to challenge with influenza virus or procedures related or influenza challenge study. For example:

    * Subject is not sero-suitable.
    * Immunocompromised status or diagnosis of active autoimmune disease.
    * Known allergy to constituents of challenge virus.
    * History of severe illness during adulthood due to a respiratory virus.
    * Inability to tolerate repeated nasopharyngeal swabs.
    * Abnormal pulmonary function in the opinion of the Investigator, as evidenced by the responses to the respiratory screening questions and /or clinically significant abnormalities in spirometry.
    * Significant history of asthma.
    * Any significant abnormality altering the anatomy of the nose or nasopharynx.
    * Any clinically significant history of epistaxis.
    * Any nasal or sinus surgery within six months of inoculation.
    * Health care workers who are reasonably likely to come into contact with severely immuno-compromised patients
    * Presence of household member or close contact who has known immunodeficiency, is receiving immunosuppressant medication, is undergoing or soon to undergo cancer chemotherapy, has been diagnosed with emphysema, COPD, or other severe lung disease, has received a bone marrow or solid organ transplant, resides in a nursing home
    * Evidence of vaccinations within the four weeks prior to inoculation/dosing, whichever occurs first.
    * Intention to receive any vaccination(s) before the Day 28 Follow Up Visit
    * Prior participation in another Human Viral Challenge Study in the preceding 12 months taken from the date of inoculation in the previous study to the date of expected inoculation in this study.
    * Receipt of systemic glucocorticoids or systemic antiviral drugs within six months prior to inoculation/dosing.
    * Receipt of any systemic chemotherapy agent, immunoglobulins or any other cytotoxic or immunosuppressive drugs at any time.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 152 (Actual)
Dates: Start 2015-08-31 (Actual); Primary Completion 2017-08-14 (Actual); Study Completion 2017-08-14 (Actual)

PRIMARY OUTCOMES:
Safety Data including but not limited to tabulation of adverse events, physical exam, vital signs, 12-lead ECGs and clinical lab results | Screening to Day 8 in Single Dose and Food Effect portions of the study
  Safety data including but not limited to tabulation of adverse events, physical exam, vital signs, 12-lead ECGs and clinical lab results (including chemistry, hematology, and urinalysis).
  Note that in the Multiple Ascending Dose (MAD) portion of the study, the time frame is from Screening to Day 17 (MAD) and for the Viral Challenge portion of the study the time frame is from Screening to Day 28 (Viral Challenge).
Safety Data including but not limited to tabulation of adverse events, physical exam, vital signs, 12-lead ECGs and clinical lab results | Screening to Day 17 in the Multiple Ascending Dose portion of the study
  Safety data including but not limited to tabulation of adverse events, physical exam, vital signs, 12-lead ECGs and clinical lab results (including chemistry, hematology, and urinalysis).
Safety Data including but not limited to tabulation of adverse events, physical exam, vital signs, 12-lead ECGs and clinical lab results | Screening to Day 28 in the Viral Challenge portion of the study.
  Safety data including but not limited to tabulation of adverse events, physical exam, vital signs, 12-lead ECGs and clinical lab results (including chemistry, hematology, and urinalysis).

SECONDARY OUTCOMES:
Cmax: AL-794 | From baseline to Day 8 for Single Dose and Food Effect cohorts
  Pharmacokinetic parameter of ALS-033719 and ALS-033927 (and other metabolites, if applicable) in plasma following single dose administration
Cmax: AL-794 | From baseline to Day 17 for Multiple Ascending Dose Cohorts
  Pharmacokinetic parameter of ALS-033719 and ALS-033927 (and other metabolites, if applicable) in plasma following multiple dose administration
AUC: AL-794 | From baseline to Day 8 for Single Dose and Food Effect cohorts
  Pharmacokinetic parameter of ALS-033719 and ALS-033927 (and other metabolites, if applicable) in plasma following single dose administration
AUC: AL-794 | From baseline to Day 17 for Multiple Ascending Dose cohorts
  Pharmacokinetic parameter of ALS-033719 and ALS-033927 (and other metabolites, if applicable) in plasma following multiple dose administration
CMax: Fed vs. Fasted | First dose to Day 8 (Single Ascending Dose/Food Effect)
  Comparison of Cmax after a single oral dose in HV in fasted conditions as compared with fed conditions.
AUC: Fed vs. Fasted | First dose to Day 8 (Single Ascending Dose/Food Effect)
  Comparison of AUC after a single oral dose in HV in fasted conditions as compared with fed conditions.
Influenza Viral Load | Baseline to Day 28
  AUC0-t of influenza viral load, as determined by quantitative polymerase chain reaction (PCR) assay of nasopharyngeal swab, from baseline (i.e., immediately prior to treatment onset) through checkout, Day 17, and completion of study
Peak influenza viral load after treatment | inoculation to Day 28
  Peak influenza viral load after treatment onset, as determined by quantitative PCR assay of nasopharyngeal swab

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm Boyce, Principal Investigator — HMR
Locations (1):
- Hammersmith Medicines Research Ltd (HMR), London, United Kingdom

REFERENCES:
- [Derived] Yogaratnam J, Rito J, Kakuda TN, Fennema H, Gupta K, Jekle CA, Mitchell T, Boyce M, Sahgal O, Balaratnam G, Chanda S, Van Remoortere P, Symons JA, Fry J. Antiviral Activity, Safety, and Pharmacokinetics of AL-794, a Novel Oral Influenza Endonuclease Inhibitor: Results of an Influenza Human Challenge Study. J Infect Dis. 2019 Jan 7;219(2):177-185. doi: 10.1093/infdis/jiy410. PMID 30053042
- [Derived] Kakuda TN, Yogaratnam J, Rito J, Boyce M, Mitchell T, Gupta K, Symons JA, Chanda S, Van Remoortere P, Fry J. Phase I study on safety and pharmacokinetics of a novel influenza endonuclease inhibitor, AL-794 (JNJ-64155806), following single- and multiple-ascending doses in healthy adults. Antivir Ther. 2018;23(7):555-566. doi: 10.3851/IMP3244. Epub 2018 Jun 21. PMID 29927386